CLINICAL TRIAL: NCT01250925
Title: Effect of Contact Lens Wear on Immune Cell Density and Morphology of the Ocular Surface: A Laser In Vivo Confocal Microscopy Study
Brief Title: Effect of Contact Lens Wear on Immune Cell Density and Morphology of the Ocular Surface
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Collaborators: University of Iowa (Other); Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 10-04-029
Record Dates: First submitted 2010-11-29; First posted 2010-12-01 (Estimated); Results first posted 2017-01-10 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2013-04

CONDITIONS: Myopia; Refractive Error
Keywords: Contact lens; Lens care
MeSH Terms: conditions — Myopia; Refractive Errors

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- OPTI-FREE® RepleniSH® (Active Comparator): 33 participants will be assigned to use this lens care regimen during the six-week assessment period
  Interventions: Drug: OPTI-FREE® RepleniSH®
- Clear Care® (Active Comparator): 33 participants will be assigned to use this lens care regimen during the six-week assessment period
  Interventions: Drug: Clear Care®
- ReNu MultiPlus® MultiPurpose Solution (Active Comparator): 33 participants will be assigned to use this lens care regimen during the six-week assessment period
  Interventions: Drug: ReNu MultiPlus® MultiPurpose Solution

INTERVENTIONS:
Drug: ReNu MultiPlus® MultiPurpose Solution — Contact lens care regimen
  Arms: ReNu MultiPlus® MultiPurpose Solution
Drug: OPTI-FREE® RepleniSH® — Contact Lens care regimen
  Arms: OPTI-FREE® RepleniSH®
Drug: Clear Care® — Contact lens care regimen
  Arms: Clear Care®

SUMMARY:
The purpose of this study is to utilize in-vivo confocal microscopy to describe differences in corneal epithelial immune status across three lens care regimens in new contact lens wearers.

DETAILED DESCRIPTION:
An estimated 40 million people in the United States wear contact lenses, with approximately 38 million soft lens wearers and 2 million rigid gas permeable lens wearers. The ocular surface has been shown to respond to the introduction of foreign materials with upregulation of proinflammatory mediators, leading to an increase in inflammation. The corneal can show a foreign body immune response to contact lenses. The purpose of this study is to utilize in-vivo confocal microscopy to describe differences in corneal epithelial immune status across the three lens care regimens in new contact lens wearers.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be 18 years of age and may be of any race and either gender.
2. Subjects must not have ever worn contact lenses.
3. Subjects must have normal, healthy eyes.

Exclusion Criteria:

1. Subjects must not use additional lens cleaners.
2. subjects must not have any ocular or systemic disease.
3. Subjects must not have history of ocular surgery/trauma within the last 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2010-08; Primary Completion 2012-02 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pedram Hamrah, MD, Principal Investigator — Massachusetts Eye and Ear Infirmary; Christine Sindt, OD, Principal Investigator — University of Iowa
Locations (2):
- United States (2):
  - University of Iowa, Iowa City, Iowa
  - Massachusetts Eye and Ear Infirmary, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 94 Neophyte contact lens wearers were fitted for one of 3 types of contact lenses (Bausch and Lomb PureVision; Vistakon Acuvue Oasys or Cooper Vision Biofinity) and were then randomized into one of three test articles (care regimens): OptiFree RepleniSH Multi-Purpose Disinfecting Solution, Clear Care or ReNu MultiPlus Multi-Purpose Solution.
Pre-assignment Details: 127 subjects were screened, out of which 94 were successfully enrolled and 35 were screenfailed due to non-normal clinical findings. Of the enrolled, 10 did not complete the study visits.
Period: Overall Study
Arm/Group | OPTI-FREE® RepleniSH® | Clear Care® | ReNu MultiPlus® MultiPurpose Solution
Started | 31 | 31 | 32
Completed | 26 | 28 | 30
Not Completed | 5 | 3 | 2
Not completed — Lost to Follow-up | 1 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0
Not completed — Protocol Violation | 2 | 0 | 0
Not completed — Physician Decision | 0 | 2 | 1
Not completed — Adverse Event | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OPTI-FREE® RepleniSH® | Clear Care® | ReNu MultiPlus® MultiPurpose Solution | Total
Number analyzed (Participants) | 31 | 31 | 32 | 94
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 31 | 31 | 32 | 94
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.7 (10.3) | 32.9 (12.2) | 30.6 (9.1) | 31.4 (10.5)
Gender [Count of Participants; unit: Participants]
  Female | 23 | 18 | 14 | 55
  Male | 8 | 13 | 18 | 39
Region of Enrollment [Number; unit: participants]
  United States | 31 | 31 | 32 | 94

OUTCOME MEASURES:

1. Primary Outcome: Corneal Epithelial Immune Dendritic Cell Density (Central Cornea)
Description: The primary statistical objective is to describe differences in efficacy between regimens, specifically for measures of epithelial immune status. Immune status will be assessed via density of dendritic and non-dendritic immune cells.
Time Frame: Six weeks
Population: Participants who completed all visits were analyzed.
Measure: Mean (Standard Error); unit: cells/mm2
Units Other Than Participants: eyes
Arm/Group | OPTI-FREE® RepleniSH® | Clear Care® | ReNu MultiPlus® MultiPurpose Solution
Number analyzed (Participants) | 26 | 28 | 30
Number analyzed (eyes) | 52 | 56 | 60
cells/mm2 | 46.2 (9.4) | 44.8 (11.6) | 62.3 (12.2)

2. Secondary Outcome: Number of Participants With Slit-lamp Findings, Corrected Visual Acuity (Snellen) and Adverse Events
Description: The safety analysis will be based on slit-lamp findings, corrected visual acuity (Snellen) and adverse events (if any). No inferential statistical analyses are planned for any safety variable.
Time Frame: Six weeks
Population: Participants who completed the study visits were analyzed.
Measure: Number; unit: participants
Units Other Than Participants: eyes
Arm/Group | OPTI-FREE® RepleniSH® | Clear Care® | ReNu MultiPlus® MultiPurpose Solution
Number analyzed (Participants) | 26 | 28 | 30
Number analyzed (eyes) | 52 | 56 | 60
participants | 0 | 1 | 1

3. Primary Outcome: Corneal Epithelial Immune Dendritic Cell Density (Inferior Cornea)
Description: as for outcome 1
Time Frame: Six weeks
Population: Participants who completed the study visits were analyzed.
Measure: Mean (Standard Error); unit: cells/mm2
Units Other Than Participants: eyes
Arm/Group | OPTI-FREE® RepleniSH® | Clear Care® | ReNu MultiPlus® MultiPurpose Solution
Number analyzed (Participants) | 26 | 28 | 30
Number analyzed (eyes) | 52 | 56 | 60
cells/mm2 | 109.0 (12.2) | 90.1 (9.7) | 113.6 (9.3)

4. Primary Outcome: Corneal Epithelial Immune Dendritic Cell Density (Nasal Cornea)
Description: as for outcome 1
Time Frame: Six weeks
Population: Participants who completed the study visits were analyzed.
Measure: Mean (Standard Error); unit: cells/mm2
Units Other Than Participants: eyes
Arm/Group | OPTI-FREE® RepleniSH® | Clear Care® | ReNu MultiPlus® MultiPurpose Solution
Number analyzed (Participants) | 26 | 28 | 30
Number analyzed (eyes) | 52 | 56 | 60
cells/mm2 | 77.7 (8.6) | 67.8 (8.1) | 73.6 (6.6)

5. Primary Outcome: Corneal Epithelial Immune Dendritic Cell Density (Superior Cornea)
Description: as for outcome 1
Time Frame: Six weeks
Population: Participants who completed the study visits were analyzed.
Measure: Mean (Standard Error); unit: cells/mm2
Units Other Than Participants: eyes
Arm/Group | OPTI-FREE® RepleniSH® | Clear Care® | ReNu MultiPlus® MultiPurpose Solution
Number analyzed (Participants) | 26 | 28 | 30
Number analyzed (eyes) | 52 | 56 | 60
cells/mm2 | 106.1 (15.2) | 92.5 (9.3) | 106.1 (11.3)

6. Primary Outcome: Corneal Epithelial Immune Dendritic Cell Density (Temporal Cornea)
Description: as for outcome 1
Time Frame: Six weeks
Population: Participants who completed the study visits were analyzed.
Measure: Mean (Standard Error); unit: cells/mm2
Units Other Than Participants: eyes
Arm/Group | OPTI-FREE® RepleniSH® | Clear Care® | ReNu MultiPlus® MultiPurpose Solution
Number analyzed (Participants) | 26 | 28 | 30
Number analyzed (eyes) | 52 | 56 | 60
cells/mm2 | 63.2 (12.2) | 59.0 (8.8) | 58.7 (5.7)

7. Primary Outcome: Corneal Epithelial Immune Non-Dendritic Cell Density (Central Cornea)
Description: as for outcome 1
Time Frame: Six weeks
Population: Participants who completed all visits were analyzed.
Measure: Mean (Standard Error); unit: cells/mm2
Units Other Than Participants: eyes
Arm/Group | OPTI-FREE® RepleniSH® | Clear Care® | ReNu MultiPlus® MultiPurpose Solution
Number analyzed (Participants) | 26 | 28 | 30
Number analyzed (eyes) | 52 | 56 | 60
cells/mm2 | 0.3 (0.2) | 0.4 (0.2) | 0.4 (0.2)

8. Primary Outcome: Corneal Epithelial Immune Non-Dendritic Cell Density (Inferior Cornea)
Description: as for outcome 1
Time Frame: Six weeks
Population: Participants who completed all visits were analyzed.
Measure: Mean (Standard Error); unit: cells/mm2
Units Other Than Participants: eyes
Arm/Group | OPTI-FREE® RepleniSH® | Clear Care® | ReNu MultiPlus® MultiPurpose Solution
Number analyzed (Participants) | 26 | 28 | 30
Number analyzed (eyes) | 52 | 56 | 60
cells/mm2 | 0.4 (0.2) | 0.5 (0.2) | 0.7 (0.4)

9. Primary Outcome: Corneal Epithelial Immune Non-Dendritic Cell Density (Nasal Cornea)
Description: as for outcome 1
Time Frame: Six weeks
Population: Participants who completed all visits were analyzed.
Measure: Mean (Standard Error); unit: cells/mm2
Units Other Than Participants: eyes
Arm/Group | OPTI-FREE® RepleniSH® | Clear Care® | ReNu MultiPlus® MultiPurpose Solution
Number analyzed (Participants) | 26 | 28 | 30
Number analyzed (eyes) | 52 | 56 | 60
cells/mm2 | 1.6 (0.9) | 1.2 (0.5) | 1.1 (0.5)

10. Primary Outcome: Corneal Epithelial Immune Non-Dendritic Cell Density (Superior Cornea)
Description: as for outcome 1
Time Frame: Six weeks
Population: Participants who completed all visits were analyzed.
Measure: Mean (Standard Error); unit: cells/mm2
Units Other Than Participants: eyes
Arm/Group | OPTI-FREE® RepleniSH® | Clear Care® | ReNu MultiPlus® MultiPurpose Solution
Number analyzed (Participants) | 26 | 28 | 30
Number analyzed (eyes) | 52 | 56 | 60
cells/mm2 | 0.2 (0.1) | 0.6 (0.2) | 0.3 (0.2)

11. Primary Outcome: Corneal Epithelial Immune Non-Dendritic Cell Density (Temporal Cornea)
Description: as for outcome 1
Time Frame: Six weeks
Population: Participants who completed all visits were analyzed.
Measure: Mean (Standard Error); unit: cells/mm2
Units Other Than Participants: eyes
Arm/Group | OPTI-FREE® RepleniSH® | Clear Care® | ReNu MultiPlus® MultiPurpose Solution
Number analyzed (Participants) | 26 | 28 | 30
Number analyzed (eyes) | 52 | 56 | 60
cells/mm2 | 0.4 (0.2) | 0.7 (0.3) | 0.8 (0.5)

ADVERSE EVENTS:
Time Frame: Six weeks
Arm/Group | OPTI-FREE® RepleniSH® | Clear Care® | ReNu MultiPlus® MultiPurpose Solution
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/31 | 0/32
Other Adverse Events (participants affected / at risk) | 0/31 | 1/31 | 1/32
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OPTI-FREE® RepleniSH® (N=31) | Clear Care® (N=31) | ReNu MultiPlus® MultiPurpose Solution (N=32)
Eye irritation (Eye disorders) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less